CLINICAL TRIAL: NCT05231278
Title: Needle-Based Confocal Laser Endomicroscopy to Aid in Lung Nodule Localization by Robotic-Assisted Navigational Bronchoscopy
Brief Title: Confocal Laser Endomicroscopy Nodule Localization by Robotic Bronchoscopy
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JJEI202101
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lung Neoplasms
Keywords: Peripheral pulmonary nodule; Needle-based confocal laser endomicroscopy; Robotic-assisted bronchoscopy; Monarch
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- nCLE aided RANB biopsy (Experimental): Single arm study
  Interventions: Device: nCLE aided RANB biospy

INTERVENTIONS:
Device: nCLE aided RANB biospy — nCLE aided RANB biopsy procedure using the Monarch® robotic-assisted navigational bronchoscopy platform and Cellvizio® I.V.E. system with AQ-Flex™ 19 Confocal Miniprobe™ used in combination with Fluorescein.

SUMMARY:
This study is designed to evaluate the safety and feasibility of real-time needle-based confocal laser endomicroscopy (nCLE) in improving diagnostic accuracy of robotic-assisted bronchoscopy (RANB) biopsy performed with the Monarch® Endoscopy Platform in patients with peripheral pulmonary nodules (PPN).

DETAILED DESCRIPTION:
Robotic-assisted navigational bronchoscopy (RANB) improves accuracy of lesion localization and diagnostic yield of the peripheral pulmonary nodule (PPN) biopsy compared to conventional flexible bronchoscopy. Needle based confocal laser endomicroscopy (nCLE) allows real-time microstructural imaging of lung nodule tissues at the needle tip. The study is designed to evaluate the safety and feasibility of utilizing nCLE during RANB biopsy procedure to optimize needle position and diagnostic accuracy, as well as reduce or replace the need for additional imaging tools such as radial endobronchial ultrasound (r-EBUS), cone beam computed tomography (CBCT), and/or fluoroscopy during RANB biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years at signing of informed consent form (ICF).
* Undergoing standard-of-care RANB for a solid lung nodule, which is considered to be at intermediate- to high-risk for malignancy as determined by the investigator per the institution's standard of care.
* ICF signed before any study procedures are initiated.

Exclusion Criteria:

* Medical contraindication to bronchoscopy under general anesthesia, or lack of physical fitness to undergo bronchoscopy under general anesthesia or to follow the study processes, as assessed by the investigator.
* Presence of uncorrectable bleeding disorders, or anticoagulation/anti-platelet aggregation therapy that cannot be withheld for an appropriate interval prior to the procedure, as defined per the institution's standard of care.
* Medical devices interfering with electro-magnetic navigation, including but not limited to pacemakers.
* Subjects who have a target lesion that shows endobronchial involvement on chest CT.
* Participation in any other clinical trial within 30 days of enrollment, that would interfere with this study.
* Known hypersensitivity to fluorescein sodium or any other ingredients in the fluorescein product.
* Planned surgical resection at the time of bronchoscopy
* Female subjects who are pregnant or nursing at the time of the procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
'Tool-in-lesion' positioning accuracy of nCLE during RANB biopsy. | Intra-procedure
  The accuracy of the positional relationship between the nCLE needle/probe and the index PPN will be determined using CBCT imaging.

SECONDARY OUTCOMES:
Sensitivity of the real-time nCLE imaging assessment for malignancy | Intra-procedure
  The real-time nCLE imaging assessment of the index PPN for malignancy will be compared to the histopathology biopsy results of the index PPN.
Diagnostic yield | up to 12 months post procedure
  Diagnostic yield for all nCLE aided RANB biopsy performed for the index PPN will be evaluated based on histopathological assessment of acquired tissue samples.
Sensitivity of the post-procedure nCLE image assessment for malignancy | Intra-procedure
  The post-procedure nCLE image assessment of the index PPN for malignancy will be compared to the histopathology biopsy results of the index PPN.
Intra- and inter-observer agreement of the post-procedure nCLE imaging for malignancy | Intra-procedure
  The post-procedure nCLE image assessment of the index PPN will be obtained by multiple independent, blinded raters; the intra- and interobserver agreement will be determined.
Safety of nCLE aided RANB biopsy procedure | up to 30 days post procedure
  The safety of nCLE aided RANB biopsy procedure will be reported as the number and frequency of adverse events (AEs) and procedure-related AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Balaji Laxmanan, MD, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (4):
- United States (4):
  - John Muir Health, Concord, California
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center of the American Oncologic Hospital, Inc., Philadelphia, Pennsylvania